CLINICAL TRIAL: NCT06716398
Title: A Randomized Investigator-blinded Comparative Study to Assess the Efficacy of the Cosmetic Care Product RV4133C - Formula JT2559 in Subjects With Facial Acne, During a 3-month-associated-treatment Phase Followed by a 3-month-maintenance Phase
Brief Title: A Comparative Study of Cosmetic Product in Subjects With Facial Acne During an Associated-treatment Phase Followed by a Maintenance Phase
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RV4133C20230380
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Acne
Keywords: acne; face; young adults; teenagers; treatment phase; maintenance
MeSH Terms: conditions — Acne Vulgaris; Facies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental)
  Interventions: Other: Test product
- Comparative group (Placebo Comparator)
  Interventions: Other: Comparator product

INTERVENTIONS:
Other: Test product — Twice daily applications, in association of a reference medical treatment during a 3-month-associated-treatment phase, then alone during a 3-month-maintenance phase. The product is applied to the entire face.
  Arms: Test Group
Other: Comparator product — Twice daily applications, in association of a reference medical treatment during a 3-month-associated-treatment phase, then alone during a 3-month-maintenance phase. The product is applied to the entire face.
  Arms: Comparative group

SUMMARY:
In this study, we are interested in the global benefit of the tested product as complementary care to a topical medical treatment during a 3 month-associated treatment phase followed by a 3 month-maintenance phase, compared to a light moisturizing cream, in teenagers and adults with acne. We also want to evaluate the tolerance of the tested product in association and in maintenance of the topical medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged between 14 and 24 years (included)
* Subject with facial acne with score index severity IGA = 2 or 3, assessed on a scale ranged from 0 to 4.
* Subject for whom a prescription of 12 weeks of a reference topical medical treatment is required from the day of the inclusion visit, for mild to moderate face acne

Exclusion Criteria:

Criteria related to the disease:

* Facial skin disease other than acne, skin abnormalities, or dermatological condition on the face liable to interfere with the study assessments
* Acne conglobata, Acne fulminans, nodulocystic acne or acneiform eruptions, according to investigator's assessment
* Other type of pigmentation disorder than acne-related PIH liable to interfere with the study assessments according to the investigator

Criteria related to treatments and/or products:

- Topical or oral treatment established or modified during the previous weeks or planned to be established or modified during the study, liable to interfere with the evaluation of the efficacy or cutaneous tolerance of the investigational products

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of number of total acne lesions on the face | Assessment after 24 weeks of use
  Number of total acne lesions by counting according to the Lucky method performed by the investigator

SECONDARY OUTCOMES:
Investigator's global assessment (IGA) | Assessment at baseline and after 4 weeks, 12 weeks, 16 weeks and 24 weeks of use
  Assessed by the investigator on the face on a 5-point scale ranged from 0 (clear) to 4 (severe)
Acne lesions counting | Assessment at baseline and 1 week, 4 weeks, 12 weeks, 16 weeks and 24 weeks of use
  Number of all type of acne lesions by counting according to subject's photographs analysis using acne Artificial Intelligence
Acne QoL questionnaire | Assessment at baseline and after 4 weeks, 12 weeks, 16 weeks and 24 weeks of use
  Assessed by the subject via a specific questionnaire of 19 questions
Subject's Global change Assessment (SGA) | Assessment after 4 weeks, 12 weeks, 16 weeks and 24 weeks of use
  Assessed by the subject via a 7-point scale: SGA of acne severity
Post-Inflammatory Hyperpigmentation (PIH) lesions counting | Assessment at baseline and after 4 weeks, 12 weeks, 16 weeks and 24 weeks of use
  Number of PIH lesions by counting according to the Lucky method performed by the investigator
Post-Inflammatory Erythema (PIE) lesions counting | Assessment at baseline and after 4 weeks, 12 weeks, 16 weeks and 24 weeks of use
  Number of PIE lesions by counting according to the Lucky method performed by the investigator
Subject's Global change Assessment (SGA) of post inflammatory lesions | Assessment at baseline and after 4 weeks, 12 weeks, 16 weeks and 24 weeks of use
  Assessed by the subject via a 7-point scale: SGA of post inflammatory lesions (PIH and PIE)
Acne worsening/ relapse | Assessment after 4 weeks, 12 weeks, 16 weeks and 24 weeks of use
  Number and percentage of acne worsening/ relapse, defined by the investigator by the necessity to change the topical medical treatment and/ or to introduce an oral medical treatment for facial acne
Time to relapse | Assessment after 4 weeks and 12 weeks of use, without reference medical treatment
  The time to first acne relapse will be calculated from the date of Visit 3 (start of maintenance phase) to the date of failure (acne relapse).
Global tolerance assessed by the investigator on a 5-point scale | Assessment after 4 weeks, 12 weeks, 16 weeks and 24 weeks of use
Compliance of the subjects to the product RV4133C | Through study completion, 6 months
  The subject will report his/her compliance in a subject's diary
Cosmetic satisfaction as regards to the use of the test product RV4133C by Cosmetic acceptability questionnaire assessed by the patient | Assessed after 4 weeks of use
  A questionnaire with a scale from 0 to 10 responding to statements about the effect of the product (0=not at all agree, 10=completely agree).

CONTACTS AND LOCATIONS:
Locations (1):
- UNIFESP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No